CLINICAL TRIAL: NCT01631591
Title: Prevalence of Food Allergies in a Cohort of Adult Patients With Eosinophilic Esophagitis
Acronym: EE
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Richard F. Lockey, MD, Division Director, Prinicpal Investogator, University of South Florida
Other Study IDs: eosinophilic esophagitis
Record Dates: First submitted 2012-06-27; First posted 2012-06-29 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Eosinophilic Esophagitis; Food Allergies
MeSH Terms: conditions — Eosinophilic Esophagitis; Food Hypersensitivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- eosinophilic esophagitis: PATIENTS WITH A CURRENT DIAGNOSIS OF eosinophilic esophagitis.
- GERD: PATIENTS WITH A DIAGNOSIS WITH GERD.

SUMMARY:
Eosinophilic esophagitis is characterized by an eosinophilic infiltration of the esophagus. It presents clinically with a variety of symptoms including dysphagia, emesis, and food impaction. Although the underlying mechanism is different, gastroesophageal reflux can present with similar clinical findings but can be distinguished from eosinophilic esophagitis by the number of eosinophils present on esophageal biopsy. In children, food allergies play a role in exacerbating eosinophilic esophagitis, but the role of food allergies in adults is uncertain. In this study, we aim to determine the prevalence of food allergies in a cohort of adults with eosinophilic esophagitis.

DETAILED DESCRIPTION:
Study Population Male and female subjects, ages 18 years and older with findings of > 15 eosinophils per high powered field by endoscopic esophageal biopsy. Patients should also have symptoms consistent with eosinophilic esophagitis including dysphagia, heartburn, epigastric pain, recurrent vomiting, or food impaction. The comparative group will include male and female subjects, ages 18 years and older with a previous diagnosis of gastroesophageal reflux with findings of < 15 eosinophils per high power field by endoscopic esophageal biopsy.

Inclusion Criteria

1. Male and female subjects 18 years and older
2. Previous diagnosis of eosinophilic esophagitis with clinical symptoms including heartburn, dysphagia, vomiting, epigastric pain, recurrent vomiting, food impaction as well > 15 eosinophils per high powered field (400x magnification) by endoscopic esophageal biopsy in both the proximal and distal esophagus
3. Previous diagnosis of gastroesophageal reflux with < 15 eosinophils per high powered field (400x magnification) by endoscopic biopsy

Exclusion Criteria

1. Male and female subjects less than 18 years of age
2. Pregnant female subjects
3. Subjects who are receiving systemic steroids and are unable to stop prior to enrollment
4. Subjects who are receiving systemic antihistamines and are unable to stop prior to enrollment
5. Subjects who are unable to cooperate/comply with study procedures or communicate with investigator in order to successfully complete the study
6. Subjects with severe skin disorders such as atopic dermatitis, dermatographism, or psoriasis who would be unable to complete skin or patch testing
7. Subjects with an infirmity, disability, or geographical location which seems likely to prevent regular attendance for patient visit Risks Skin testing with prick methodology has a risk of systemic reaction of less than 0.1% per 40 tests, however, no deaths have been reported with this method of testing. Systemic reactions are readily treated using Injectable epinephrine with oral antihistamines and oral corticosteroids (prednisone). Patch testing has no known associated risk for development of systemic reactions. Phlebotomy is associated with a minimal risk of bleeding, significant local discomfort, and infection from the needle puncture.

Benefits Treatment options for adults with eosinophilic esophagitis are limited. Food allergies are a known contributor to this disorder in children and a better understanding of food allergies in adult subjects may provide additional treatment options.

Adverse Events and Withdrawal Criteria All subjects will be assessed for adverse events at each study visit. If any adverse events are experienced by the subject, the investigator will document the event within the subject's file and promptly report the event to the IRB. The investigators involved with this study will determine if a participant needs to be withdrawn from the study based upon the subject's health and medical history.

Sample Size Sample size estimation is based on the assumption that up to 50% of adults with eosinophilic esophagitis (EE) will have a positive skin test to food and 10% of adults without EE will have a positive skin test to food. With this assumption, a total of 40 subjects are needed, 20 per group, in order to achieve at least 80% power with two sided test at alpha level of 0.05 and beta 0.2.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects 18 years and older
2. Previous diagnosis of eosinophilic esophagitis with clinical symptoms including heartburn, dysphagia, vomiting, epigastric pain, recurrent vomiting, food impaction as well > 15 eosinophils per high powered field (400x magnification) by endoscopic esophageal biopsy in both the proximal and distal esophagus
3. Previous diagnosis of gastroesophageal reflux with < 15 eosinophils per high powered field (400x magnification) by endoscopic biopsy

Exclusion Criteria:

1. Male and female subjects less than 18 years of age 2. Pregnant female subjects 3. Subjects who are receiving systemic steroids and are unable to stop prior to enrollment 4. Subjects who are receiving systemic antihistamines and are unable to stop prior to enrollment 5. Subjects who are unable to cooperate/comply with study procedures or communicate with investigator in order to successfully complete the study 6. Subjects with severe skin disorders such as atopic dermatitis, dermatographism, or psoriasis who would be unable to complete skin or patch testing 7. Subjects with an infirmity, disability, or geographical location which seems likely to prevent regular attendance for patient visit

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects, ages 18 years and older with findings of > 15 eosinophils per high powered field by endoscopic esophageal biopsy. Patients should also have symptoms consistent with eosinophilic esophagitis including dysphagia, heartburn, epigastric pain, recurrent vomiting, or food impaction. The comparative group will include male and female subjects, ages 18 years and older with a previous diagnosis of gastroesophageal reflux with findings of < 15 eosinophils per high power field by endoscopic esophageal biopsy.
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2011-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of food allergies in a cohort of adult patients with EE. | Study to close on or around May 2014

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida, Tampa, Florida, United States